CLINICAL TRIAL: NCT06008145
Title: COPD Case Finding In Nottingham and District: C-FIND COPD A Pilot Study
Acronym: C-FIND
Status: Active, not recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 23RM005
Record Dates: First submitted 2023-07-20; First posted 2023-08-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and nasal brush
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Targeted Lung Health Check (TLHC) is currently being rolled out in many regions of the United Kingdom and has just started in Nottingham. The same cohort of people are also at high risk for Chronic Obstructive Pulmonary Disease (COPD), a lung condition often caused by smoking and leading to breathlessness and cough. This study aims to provide pilot evidence of the role of breathing tests in those who have had a Computerised Tomography (CT) scan, in order to early diagnose COPD. Currently, at diagnosis, many patients have lost 30-40% of lung function already, which is not reversible.

This study will use the Nottingham University Hospitals Trust Mobile Research Unit. The unit will follow the CT scanner route 2-3 weeks later, and people who have had a CT scan will be invited for breathing tests. Participants will also collect further information on potential treatment options for people diagnosed with COPD earlier -including smoking cessation, symptom management and general health advice (vaccinations, diet, activity and managing infections). There is also an optional blood test.

The study aims are to determine the uptake and acceptability of breathing tests in patients at high risk of COPD, and if a community based approach co-locating with TLHC can increase uptake.

A qualitative sub-study has been added to assess the opportunities or barriers for people being invited for a COPD diagnosis visit in the community. This sub-study will have a recruitment target of 20 participants. It will involve transcribed interviews. This will help determine the accessibility of the mobile research unit in use for this study.

DETAILED DESCRIPTION:
Ever smokers, aged between 55 to 74 years are invited for a telephone risk assessment. Those who are high risk (based on validated lung cancer risk scores, which incorporate a number of variables, including age and smoking intensity) are then sequentially invited for a CT scan in a certain locality of Nottingham as part of the TLHC. As the programme is introduced the number of invites per month will increase from 500 to 1800. It is anticipated that 40 to 45% of those will take up the invite and have a CT scan. At the time of their CT scan all smokers will be offered smoking cessation.

The clinical pathway incorporates that the CT scans will be reported by Heart Lung Health , with responsible clinician - Dr O'Dowd. Patients identified as having cancer or high likelihood will be approached and commenced on a cancer diagnostic pathway. This study addresses people who are not entering this pathway.

Two-three weeks after the CT scan, the clinical team will invite people to attend for a research study to assess lung health if they have symptoms of cough, breathlessness or 2 or more courses antibiotics in the last 15 months. No further reminder will be sent. The investigators will not excluding people with COPD already and will not turn away high-risk people who self-present even if not had a CT.

The invite will include mention of when the mobile unit is open and in their locality, what the visit consists of and that participants are free to come down at a convenient time. A telephone number and e-mail will be provided if somebody contacts the investigators and would prefer to be seen in a standard research unit - an appointment will be provided. The letter will remind participants that this cannot cover broader medical issues or emergencies, where usual clinical advice should be sought.

Following informed consent, the following will occur by trained clinical research practitioners and under the support of a research nurse.

* Questionnaires:

  * Symptom scores and information on tobacco smoking / other exposures, past medical history, medication
  * COPD Assessment Test (CAT) Quality of Life score
  * Medical Research Council (MRC) breathlessness score
  * Exacerbation frequency
  * EQ5D - Health Status
* Observations:

  * Oximetry for heart rate and oxygen saturations
  * Height
  * Weight
  * Blood pressure
* Postbronchodilator spirometry - salbutamol delivered by trained staff.
* Forced Oscillation Technique (FOT)- a non-clinically used breathing test but might have a role in early detection.
* Approach for future research and store research data obtained here / review medical records for future medicines.
* Invite to provide a blood sample and nasal swab for early markers of COPD - optional and currently of no clinical relevance.

Those with clinical evidence of COPD will be given information by a registered Health Care professional trained to do so on:

* COPD and what it is.
* Need for immunisations.
* General health education, self-management and tobacco cessation where indicated.
* Whether further review at the surgery is required.
* Clinical information will be fed back to primary care surgery and uploaded onto medical health records, such as SystemOne. The participant will have consented to this.

The investigators will seek feedback from participants and subsequently from the primary care clinicians.

A qualitative sub-study has been added to assess the opportunities or barriers for people being invited for a COPD diagnosis visit in the community. This sub-study will have a recruitment target of 20 participants. It will involve transcribed interviews. This will help determine the accessibility of the mobile research unit in use for this study.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history - either compatible with TLHC (current or ex-smoker who are high risk based on lung cancer risk scores) or if self-presenting >10 pack years (current or ex)
* Able to provide full informed consent.

Exclusion Criteria:

* People currently undergoing active investigation or treatment for cancer
* Unable to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Targeted Lung Health Check (THLC) cohort are a population that are at high risk for COPD, a lung condition often caused by smoking. This same population will be invited to undertake breathing test in order to early diagnose COPD.
Sampling Method: Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of people who take up the invite to attend for a C-FIND visit. | 1.5 years
  0-100%

SECONDARY OUTCOMES:
Proportion diagnosed with COPD | 1.5 years
  0-100%
CAT COPD Quality of Life Score | 1 day
  Questionnaire. Wellbeing and daily life questions, scored 0-40 points, lower better
MRC breathlessness score | 1 day
  Questionnaire, self reported breathlessness grade 1-5, lower better
Exacerbation Frequency | 1 day
  0-12/year
EQ-5D-5L - Health Status | 1 day
  Questionnaire. Self reported health scale 0-100. Greater better
Oximetry for oxygen saturations | 1 day
  75-100% Oxygen saturation
Height | 1 day
  Participant height in metres - range 1.2-2.0m
Weight | 1 day
  participant weight in Kg - range 35-180Kg
BMI | 1 day
  12-60g/m2
Blood pressure diastolic | 1 day
  40-120mmHg
Post bronchodilator Spirometry | 1 day
  Forced Expired Volume (FEV)% - range 10-140% predicted
FOT-R (Resistance) | 1 day
  cmH2O.s/l
FOT-X (reactance) | 1 day
  cmH2O.s/l
FOT-AX (area of reactance) | 1 day
  cmH2O/L
FOT-Fres (resonant Frequency) | 1 day
  Hz
Blood pressure -systolic | 1 day
  75-230mmHg
What are the opportunities or barriers for people being invited for a COPD diagnosis visit in the community | From enrolment to the end of study
  To assess the barriers and opportunities presented by the use of the mobile research unit

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bolton, MD, PhD, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom